CLINICAL TRIAL: NCT00383227
Title: A Phase III, Clinical Trial Comparing the Immunogenicity and Safety of SmithKline Beecham Biologicals New Adjuvanted Hepatitis B Vaccine to a Double Dose of Engerix™-B, in Pre-haemodialysis/Haemodialysis Patients (>=15 Years of Age)
Brief Title: Comparison of Adjuvanted Hepatitis B Vaccine to Double Dose of Engerix™-B in Pre- /Haemodialysis Patients Aged ≥15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/032
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

INTERVENTIONS:
Biological: Hepatitis B adjuvanted vaccine

SUMMARY:
Comparison of adjuvanted hepatitis B vaccine to double dose of Engerix™-B in pre- /haemodialysis patients aged ≥15 years

ELIGIBILITY:
Inclusion Criteria:

* A male or female > = 15 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/ from the parents or guardians of the subject.
* Seronegative for anti-HBs antibodies, anti-HBc antibodies & Hepatitis B Surface antigen (HBsAg).
* If the subject was a female, she was of non-childbearing potential or, if of childbearing potential, she had to be abstinent or use adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination.
* Pre-haemodialysis patient* or a patient on haemodialysis.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine during the study period or within 30 days preceding the first dose of study vaccine.
* Previous vaccination against hepatitis B.
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within 6 weeks. Pregnant or lactating female
* Clinically abnormal ALT/AST values (> 3 times normal values)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 1999-12; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Anti-HBs seroprotection rates at Month 7.

SECONDARY OUTCOMES:
Solicited symptoms, unsolicited symptoms and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kong NC, Beran J, Kee SA, Miguel JL, Sanchez C, Bayas JM, Vilella A, Calbo-Torrecillas F, Lopez de Novales E, Srinivasa K, Stoffel M, Hoet B. A new adjuvant improves the immune response to hepatitis B vaccine in hemodialysis patients. Kidney Int. 2008 Apr;73(7):856-62. doi: 10.1038/sj.ki.5002725. Epub 2007 Dec 26. PMID 18160963
- [Background] Tong NK, Beran J, Kee SA, Miguel JL, Sanchez C, Bayas JM, Vilella A, de Juanes JR, Arrazola P, Calbo-Torrecillas F, de Novales EL, Hamtiaux V, Lievens M, Stoffel M. Immunogenicity and safety of an adjuvanted hepatitis B vaccine in pre-hemodialysis and hemodialysis patients. Kidney Int. 2005 Nov;68(5):2298-303. doi: 10.1111/j.1523-1755.2005.00689.x. PMID 16221232
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208129/032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register